CLINICAL TRIAL: NCT03447301
Title: The Effect of Daily Consumption of Extra Virgin Olive Oil on Blood Glucose Among Diabetic Patients: An Open-label Parallel Group Randomized Controlled Trial.
Brief Title: The Effect of Daily Consumption of Extra Virgin Olive Oil on Blood Glucose Among Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sulaiman AlRajhi Colleges (Other)
Collaborators: Qassim University (Other); Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SulaimanAC
Record Dates: First submitted 2018-02-18; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Saudi Arabia, Extra Virgin Olive Oil, Blood Glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extra virgin olive oil (Experimental): Extra virgin olive oil (30mL) daily
  Interventions: Dietary Supplement: Extra virgin olive oil (30mL daily)
- Control (No Intervention): No consumption of extra virgin olive oil

INTERVENTIONS:
Dietary Supplement: Extra virgin olive oil (30mL daily) — Intervention arm will take 30 mL of Extra virgin olive oil daily.
  Arms: Extra virgin olive oil

SUMMARY:
Saudi Arabia has the highest prevalence (24%) of type 2 diabetes mellitus (T2DM) among the modern nation states in the world. In addition, majority of Saudi diabetic patient do not have their blood glucose controlled. Data suggests that diet, rich in olive oil and nuts, significantly reduces fasting plasma glucose and HbA1c (glycated hemoglobin). Olive oil has been associated with weight reduction as well as improvements in lipid profile (increase in high density (HDL) and decrease in low-density lipoprotein (LDL)). No randomized controlled trial has specifically examined the effect of olive oil as a supplement on blood glucose among diabetics. The study objective is to test the effect of daily consumption (30 mL) of extra-virgin olive oil (EVOO) on HbA1c among patients with type 2 diabetes.

DETAILED DESCRIPTION:
Problem: Saudi Arabia has the highest prevalence (24%) of type 2 diabetes mellitus (T2DM) among the modern nation states in the world. In addition, majority of Saudi diabetic patient do not have their blood glucose controlled.

Significance: Data suggests that diet, rich in olive oil and nuts, significantly reduces fasting plasma glucose and HbA1c (glycated hemoglobin). Olive oil has been associated with weight reduction as well as improvements in lipid profile (increase in high density (HDL) and decrease in low-density lipoprotein (LDL)). No randomized controlled trial has specifically examined the effect of olive oil as a supplement on blood glucose among diabetics.

Objectives: To test the effect of daily consumption (30 mL) of extra-virgin olive oil (EVOO) on HbA1c among patients with type 2 diabetes.

Methods: The study design will be an open-label randomized controlled trial with 2 groups (EVOO versus no oil). The study will include 420 patients and each patient will be followed for 3 months. Group difference in HbA1c will be compared at 3 months to determine the effect of EVOO.

Implications: Dietary supplementation of EVOO could aid Saudi diabetic patients in keeping blood glucose levels controlled.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Type 2 diabetes within 10 years of enrollment
* baseline HbA1C > 7%,
* willing to supplement the diet with oil
* able to read and write

Exclusion Criteria:

* type 1 diabetes mellitus
* have gall-bladder or liver diseases or malabsorption or Crohn's disease
* have advanced heart disease
* have an aversion or allergy to olive oil
* already using olive oil daily as a dietary supplement
* morbidly obese (Body Mass Index >40 kg/m2)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-02-25 (Estimated); Primary Completion 2018-08-25 (Estimated); Study Completion 2018-12-25 (Estimated)

PRIMARY OUTCOMES:
HbA1c (glycated hemoglobin) | 3-month follow-up

SECONDARY OUTCOMES:
Fasting Plasma Glucose | 3-month follow-up
Lipid Profile | 3-month follow-up
  High-density lipoprotein (HDL), Low-density lipoprotein (LDL), HDL/LDL ratio, triglycerides (TG), Cholesterol
Weight | 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nazmus Saquib, PhD, Principal Investigator — Sulaiman Al-Rajhi Colleges
Locations (1):
- Buraidah Diabetic Center, Buraidah, Al-Qassim, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No